CLINICAL TRIAL: NCT07098039
Title: Cardio-Fit2: Impact of a Cardiac Rehabilitation Program in Patients With Cardiovascular Disease
Acronym: Cardio-Fit2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Virgen de la Luz (Other)
Collaborators: University of Castilla-La Mancha (Other)
Responsible Party: Principal Investigator, Susana Priego Jiménez, Diploma in physiotherapy, PhD in Socio-Health and Physical Activity Research from the UCLM International Doctoral School, with a distinction of OUTSTANDING CUM LAUDE., Hospital Virgen de la Luz
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: REG: 2023/PI0523
Record Dates: First submitted 2025-07-02; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Diseases (CVD); Cardiac Rehabilitation
Keywords: cardiac rehabilitation; cardiovascular diseases; wearables
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This project will have a prospective longitudinal design, specifically a randomized controlled trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Both the researchers who manage the data and include it in the database, as well as those who analyze it, will not know the intervention that the participants have received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hospital Cardiac rehabilitation (Experimental): The hospital cardiac rehabilitation group will attend the hospital 3 days a week for the same, for eight weeks.
  Interventions: Other: Hospital Cardiac Rehabilitation
- Semi-presential or hibrid group (Other): The hybrid format will consist of 4 in-person sessions (every two weeks) complemented by a home program until completing 3 sessions of the full program at home
  Interventions: Other: Semi-presential or hybrid group

INTERVENTIONS:
Other: Semi-presential or hybrid group — The hybrid format will consist of 4 in-person sessions (every two weeks) complemented by a home program until completing 3 sessions of the full program at home.
  Arms: Semi-presential or hibrid group
Other: Hospital Cardiac Rehabilitation — The hospital cardiac rehabilitation group will attend the hospital 3 days a week for the same, for eight weeks.
  Arms: Hospital Cardiac rehabilitation

SUMMARY:
Cardiovascular diseases (CVD) are the main cause of morbidity and mortality in the world, being responsible for 17.9 million deaths annually, according to the World Heart Federation (WHF), which represents a significant social and health cost both due to direct expenses derived from admissions and diagnostic-therapeutic methods, as well as indirect expenses secondary to work incapacity, disability and loss of autonomy that this generates. Although advanced diagnostic and therapeutic techniques have been incorporated in recent years in the acute phase of ischemic heart disease, interventions during hospitalization and after hospital discharge remain insufficient in terms of secondary prevention, a paradoxical fact, since increasingly, the available evidence, as well as the recommendation guidelines, focus on the modification of lifestyle habits and control of cardiovascular risk factors (CVRF), fundamental pillars of cardiac rehabilitation programs (PRC) as a preventive measure both in the appearance of new adverse events and in the reduction of disease progression and improvement of the functional capacity of the patient. Cardiac rehabilitation (CR) was defined by the World Health Organization (WHO) in the 1960s as "the set of activities necessary to ensure that heart patients have an optimal physical, mental and social condition, allowing them to occupy, by their own means, as normal a place as possible in society." The scientific evidence is more than consistent regarding the benefits that multidisciplinary CRP provides in terms of cardiovascular mortality and quality of life (QoL) of our patients and how these results are maintained despite changes in patient characteristics and risk, or the incorporation of new pharmacological treatments. Therefore, if we deprive our patients of these therapies, we are indirectly acting negatively on their cardiovascular prognosis, especially within the field of ischemic heart disease, although it is increasingly being extended to other areas of Cardiology such as heart failure (HF), pulmonary hypertension (PH), valvular disease,7 etc. So much so that it is already included in the latest clinical practice guidelines of the main scientific societies at European and American level, establishing participation in a CR program after acute coronary syndrome or coronary revascularization and those patients with HF as a "level of recommendation I evidence A"

DETAILED DESCRIPTION:
Currently, due to both the high percentage of patients with cardiovascular disease and the potential increase in sedentary lifestyle, with the geographical dispersion of some territories such as our integrated care area, it is vital to seek effective alternatives so that therapeutic exercise programs are carried out regularly, given that this sedentary attitude can increase the risk of mortality.40 This gives impetus to remote interventions such as telerehabilitation, as a useful paradigm to reduce this risk by being a set of technologies that has facilitated the application, monitoring and follow-up of physical exercise programming.

In today's technological era, the Internet of Things (IoT) paradigm has facilitated the incorporation of connected devices, such as smart tablets, motion sensors, activity trackers, and virtual reality systems, capable of monitoring physiological and behavioral variables in real time and acting on the data collected, thus enabling remote, personalized, and continuous interventions. These advances have begun to be used in healthcare and rehabilitation settings, with promising results.

In this way, an association has been evidenced between the home use of these technologies with moderate to high levels of participation in RCD and patient satisfaction with this modality; 46,47 with similar benefits in improving cardiovascular and psychological health, 48 which suggests that RCD with technological support is a viable option to monitor and even increase participation in the RC process, 46,48 especially for those patients who, due to their employment situation or geographical dispersion, do not have easy access to PRC. It should be taken into account that RCD may entail less medical supervision, control of physical exercise sessions with telemetry and monitoring, security and social interaction, but it is an alternative to achieve maintenance of physical activity levels in patients with CVD. 42 Some authors even recommend RCD in high-risk patients, given that the cardiovascular and psychological benefits that can be obtained by performing low-impact physical exercise at home are greater than the relative risk of an adverse event.

In this regard, several authors have shown that the implementation of home-based training protocols is safe and feasible for patients with low- and moderate-risk CVD; 50-53 with no significant difference in the relative risk of mortality between both CR modalities. 43 Other reviews reached similar conclusions without differentiating between total mortality, exercise capacity and QoL between the RCD and RCT groups. However, there was evidence of marginally higher levels of program completion by home-based participants.

One of the main weaknesses of the RCD is the lack of direct patient monitoring during the program. In this sense, the use of wearable devices overcomes this limitation, as it facilitates remote monitoring of patient activity, increasing accessibility to the RCP for people who would otherwise be unable to benefit from them. Furthermore, the use of these devices during the program contributes to improving adherence by allowing more precise monitoring of both exercise performance and various physiological variables that they record in real time.

The use of wearable devices in RCD programs improves patient adherence and allows for more effective monitoring of physical activity and physiological variables, resulting in greater program effectiveness compared to rehabilitation without remote monitoring.

The study will be conducted at the Virgen de la Luz Hospital in Cuenca, among patients with cardiac pathology described in the inclusion criteria, who will be enrolled in a cardiac rehabilitation program. The variables collected before and after the intervention will be analyzed and studied. Participants will be recruited throughout the project. Variables will be measured initially (inclusion in the program) and after the program ends (post-intervention).

The intervention will last 8 weeks (2 months). Both groups will receive the same exercise program, although the in-person group will attend the hospital 3 days a week for eight weeks, while the hybrid format will consist of 4 in-person sessions (every two weeks) supplemented with a home program until completing 3 sessions of the full program at home. Both groups will be monitored to measure adherence and ensure proper implementation of the program, as well as to adapt and personalize the exercise program and physical activity recommendations at all times. In this way, according to the classification of patients by number of steps (sedentary: < 5000 steps/day, not very active: 5000-7499 steps/day, somewhat active: 7500-9999 steps/day, active: 10000-12499 steps/day and very active: > 12499 steps/day),54 we will set the objective for the patient to be as active as possible, instructing them to try to increase the number of steps gradually, according to the recommendations of the guide for the prescription of physical exercise in patients with cardiovascular risk.

Likewise, patients will be monitored both with hospital telemetry, linked to the Ergoline training program, and with Polar H10 heart rate sensors during in-person sessions (in both groups), for subsequent analysis of electrocardiogram (ECG) signals.

The personalized exercise program for both groups will follow the following structure: warm-up (upper extremity mobilization, lower extremity and spine mobilization, for 10-15 minutes at an intensity of 1-2 on the modified Borg scale), strengthening exercises for large muscle groups (30-40% of 1RM for upper extremities and 50-60% of 1RM for lower extremities), abdominal muscle training, stretching, and relaxation or cool-down.

The program will be implemented with a respiratory muscle training program at 30-70% of the MIP (in the case of the inspiratory muscles) and the MEP (in the case of the expiratory muscles) in those patients whose respiratory pressure measurements have been less than 70% of the predicted value. To manage CVRF, they will receive health education sessions taught by a multidisciplinary team (urology, nursing, cardiology, physiotherapy, etc.). They will be given recommendations for daily physical activity (aerobic exercise) to complete the MIP, at an intensity of 60-85% of VO2 and 60-85% of the maximum heart rate (MHR) obtained by ergospirometry. This basic structure will be adapted for each patient with the goal of personalizing and maximizing the exercise dose (in terms of session duration, intensity, time, and type of exercise, following the FITT principle) based on the patient's progress and the level of physical activity reported by their activity trackers.

At the end of each week, personalized recommendations will be provided based on the analysis of data collected by wearable devices. These recommendations will be generated using adaptive recommendation systems that incorporate deep learning algorithms, allowing us to optimize the benefits of the cardiac rehabilitation program (CRP) and tailor it to each patient's individual needs, in line with the principles of personalized medicine. For patients in whom we also target weight loss as a control for CVRF due to obesity, we will encourage them to work daily at the point of maximum fat oxidation, or fatmax, to maximize the effect of PA on weight loss.

The exercise program will be implemented and reinforced by viewing the materials and videos recorded by the physical therapist, in order to achieve greater adherence to the program.

On the first day of the program, each patient will be given a Fitbit Inspire 3 activity tracker, which will be linked to a data-storage website to monitor each patient's program completion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 20 and 80.
2. Have suffered an acute event or have chronic cardiovascular disease with decreased/limited functional capacity.
3. Reside in the provinces of Cuenca, Toledo, or Albacete.
4. Willingness to participate voluntarily and acceptance of the conditions.
5. Must report the ability to access new technologies.

Exclusion Criteria:

1. Have a physical or mental condition that prevents participation.
2. Inability to adhere to the entire program, as reported in the initial consultation.
3. Are outside the age criteria defined above.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ergospirometry parameters and functional capacity | Baseline and up to eight weeks.
  Ergospirometry will be performed, in which the following parameters will be collected: VO2 peak (ml/Kg/min).

SECONDARY OUTCOMES:
Anthropometric data | Baseline and up to eight weeks
  Weight (Kg)
Heart rate | Baseline and up to eight weeks
  Heart rate will be measured before and after the program.
Dyspnoea | Baseline and up to eight weeks
  The patient's dyspnea, measured using the Modified Borg scale, from 0 (lower value) to 10 (highest value)
Biochemical parameters: HbA1c | Baseline and up to eight weeks
  Pre- and post-intervention tests will be requested: HbA1c
Muscle strength | Baseline and up to eight weeks
  It will be measured with a handgrip dynamometer (left and right) to measure hand grip strength.
Respiratory muscle strength | Baseline and up to eight weeks
  It will be measured by assessing respiratory pressures (maximum inspiratory pressure (MIP)
Nutritional ultrasound 1 | Baseline and up to eight weeks
  Ultrasound measurements of the rectus femoris muscle of the quadriceps will be performed to more accurately assess the morphological and functional status of the muscle.
Ultrasound measurements of subcutaneous adipose tissue | Baseline and up to eight weeks
  Ultrasound measurements of subcutaneous adipose tissue will be performed to assess fat distribution and correlate it with clinical variables. The ultrasound transducer is placed on the midline between the xiphoid process and the umbilicus. Images are taken during expiration, in a transverse plane, with a variable 4-10 cm probe, perpendicular to the skin. The image differentiates the superficial and deep layers.
Anxiety | Baseline and up to eight weeks
  It will be measured using the "HADS" scale; it is composed of two subscales: Depression and Anxiety, each with 7 items. The score for each subscale can range from 0 to 21, with each item having 4 response options, ranging from absence/minimal presence = 0 to maximum presence = 3. A higher score indicates greater severity or intensity of symptoms.
Quality of Life Questionnaire (SF-12) | Baseline and up to eight weeks
  Health-related quality of life will be assessed using the SF-12 questionnaire. This is a validated Likert-type tool (a shortened version of the SF-36). The number of response options ranges from three to six, depending on the item, and each question is assigned a score that is subsequently transformed into a scale of 0 to 100.
Pittsburgh Sleep Quality Questionnaire | Baseline and up to eight weeks
  It has a total of 19 questions, grouped into 10 items, each with a score ranging from 0 to 21. "0" indicates ease of falling asleep, and "21" indicates severe difficulty in all areas.
Mediterranean Diet Adherence Questionnaire (PREDIMED) | Baseline and up to eight weeks
  Adherence to the Mediterranean diet will be assessed using the "PREDIMED" questionnaire. This is a validated tool that assesses your level of adherence to the Mediterranean diet pattern with 14 simple questions.
Spirometric parameters: FEV1 | Baseline and up to eight weeks
  Ergospirometry will be performed, from which the following respiratory parameters will be obtained: FEV1
Analysis of Photoplethysmography signals | Baseline and up to eight weeks
  Photoplethysmography signals will be analyzed to assess the effect of PRC on cardiac dynamics.
Anthropometric data: height | Baseline and up to eight weeks
  height (cm)
BMI | Baseline and up to eight weeks
  weight and height will be combined to report BMI in kg/m ^2).
Cardiac Rehabilitation Program Satisfaction Questionnaire | up to eight weeks
  A program satisfaction questionnaire will be completed at the end of the program. This questionnaire will assess aspects related to the program, as well as the ease and usefulness of using the wearables and the exercise website and program materials to improve adherence.
Blood pressure | Baseline and up to eight weeks
  pre and post cardiopulmonary exercise test
SpO2 | Baseline and up to eight weeks
  oxygen saturation (pre and post CPET)
Biochemical parameters: cholesterol | Baseline and up to eight weeks
  cholesterol
Biochemical parameters: triglycerides | Baseline and up to eight weeks
  triglycerides
Biochemical parameters: pro-BNP | Baseline and up to eight weeks
  pro-BNP
Biochemical parameters: interleukins | Baseline and up to eight weeks
  interleukins
Respiratory muscle strength: PEM | Baseline and up to eight weeks
  It will be measured by assessing respiratory pressure maximum expiratory pressure (MEP)).
Depression | Baseline and up to eight weeks
  It will be measured using the "HADS" scale; it is composed of two subscales: Depression and Anxiety, each with 7 items. The score for each subscale can range from 0 to 21, with each item having 4 response options, ranging from absence/minimal presence = 0 to maximum presence = 3. A higher score indicates greater severity or intensity of symptoms.
Spirometric parameters: FVC | Baseline and up to eight weeks
  Ergospirometry will be performed, from which the following respiratory parameters will be obtained: FVC
Spirometric parameters: FEV1/FVC | Baseline and up to eight weeks
  Ergospirometry will be performed, from which the following respiratory parameters will be obtained: FEV1/FVC
Ultrasound measurements of visceral adipose tissue | Baseline and up to eight weeks
  Ultrasound measurements of visceral adipose tissue will be performed to assess fat distribution and correlate it with clinical variables.
  Visceral adipose tissue (Hamagawa technique) will be measured transversely, in cm. The distance from the edge of the parietal peritoneum to the linea alba on the inner surface at the junction of the two rectus abdominis muscles will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Virgen de la Luz, Cuenca, Cuenca, Spain

IPD SHARING:
Plan to Share IPD: No